CLINICAL TRIAL: NCT01943903
Title: Prospective LongitudinAl Trial of FFRct: Outcome and Resource IMpacts
Brief Title: The PLATFORM Study: Prospective LongitudinAl Trial of FFRct: Outcome and Resource IMpacts)
Acronym: PLATFORM
Status: Completed | Type: Observational
Sponsor: HeartFlow, Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CP-903-003
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort 1 - Standard of Care: Subjects will be referred for non-invasive and/or invasive testing and evaluation. Prior to treatment of each subject considered for percutaneous coronary intervention (PCI) and/or coronary artery bypass grafting (CABG), the investigator and the institution's heart team will review clinical data and results of the diagnostic tests to recommend a treatment strategy, according to the institution's standard practice. Cohort 1 of the study is an observational evaluation of resource utilization and outcomes based on standard practice for diagnosis and treatment of subjects with symptomatic suspected CAD and intermediate likelihood of obstructive CAD. Subjects will be followed for one year after enrollment.
- Cohort 2 - FFRCT-guided: Subjects will be referred for non-invasive and/or invasive testing and evaluation. Prior to treatment of subjects considered for PCI and/or CABG, the investigator and the institution's heart team will review the results of all available diagnostic tests, including cCTA and FFRCT, and will recommend a treatment strategy accordingly. FFRCT is a non-invasive method to evaluate the hemodynamic significance of coronary artery lesions. FFRCT calculates FFR from subject-specific cCTA data using computational fluid dynamics under rest and simulated maximal coronary hyperemic conditions. FFRCT values range between 0 and 1, and values ≤0.80 are considered hemodynamically (HD)-significant.

SUMMARY:
The objective of the PLATFORM Study is to compare clinical outcomes, resource utilization, and quality of life (QOL) of FFRCT-guided evaluation versus standard practice evaluation in patients with suspected CAD in order to further inform patients, health care providers, and other stakeholders about which technologies are most effective and efficient in the diagnosis of CAD

DETAILED DESCRIPTION:
The OVERALL OBJECTVE of this post-market, multicenter, longitudinal, prospective, consecutive cohort study is to compare clinical outcomes, resource utilization, and quality of life (QOL) in subjects receiving standard practice evaluation and treatment versus subjects receiving FFRCT-guided evaluation and treatment in subjects with suspected CAD in order to further inform patients, health care providers, and other stakeholders about which technologies are most effective and efficient in the diagnosis of CAD. Cohort 1 of this study will assess outcomes incorporating standard practice evaluation and Cohort 2 will assess outcomes incorporating FFRCT-guided evaluation. Each Cohort will be further delineated based upon initial presentation, whereas subjects presenting for initial non-invasive testing will be designated as Cohorts 1A and 2A; and subjects already referred for ICA will be designated as Cohorts 1B and 2B.

SPECIFIC OBJECTIVES for sequential cohort comparisons:

1. To compare the rate of ICA documenting non-obstructive coronary artery disease, clinical outcomes, and QOL following standard practice for diagnostic and treatment planning modalities in Cohort 1 versus incorporating FFRCT as the preferred test to guide further invasive management and medical treatment in Cohort 2;
2. To compare resource utilization following standard practice for diagnostic and treatment pathways in Cohort 1 versus incorporating FFRCT as the preferred test to guide further invasive management and medical treatment in Cohort 2;
3. To provide supporting data for generating new guidelines for diagnosis and prognosis of CAD with comparative analysis of the risk stratification with the Updated Diamond-Forrester risk model (UDF);
4. To provide society including patients, health care providers and other stakeholders with information about which diagnostic technologies are most effective and efficient in managing patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Providing written informed consent
* Subjects with intermediate likelihood of obstructive CAD with an Updated Diamond-Forrester (UDF) risk score 20-80% with symptomatic, suspected CAD who:
* In Cohort 1A & 2A only are scheduled to undergo initial clinically-indicated non-invasive coronary evaluation, and have not undergone non-invasive coronary evaluation, including exercise tolerance testing, stress echocardiography, SPECT or MRI, or cCTA, within the past 90 days OR ICA at any time; or
* In Cohort 1B & 2B only have been referred to invasive coronary angiography (ICA) and have not undergone ICA within the past 90 days
* Ability to undergo cCTA

Exclusion Criteria:

* Suspicion of acute coronary syndrome. Subjects experiencing unstable angina are not excluded where clinical documentation has ruled out a myocardial infarction.
* Prior, clinically documented myocardial infarction
* PCI prior to first test
* CABG prior to first test
* Contraindications for cCTA such as:
* Presence of pacemaker or internal defibrillator leads
* Atrial Fibrillation
* Known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status in women of childbearing potential
* Body mass index >35 kg/m2
* Contraindication to acute beta blockade
* Contraindication to acute sublingual nitrate administration
* Prosthetic heart valve
* Contraindications to FFRCT
* Complex Congenital Heart disease other than anomalous coronary origins alone
* Ventricular septal defect with known Qp/Qs>1.4
* Requiring an emergent procedure within 48 hours of presentation
* Evidence of active clinical instability, including cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, or NYHA Grade III or IV congestive heart failure or acute pulmonary edema
* Any active, serious, life-threatening disease with a life expectancy of less than 2 years
* Inability to comply with study follow-up requirements
* Current participation in any other clinical trial involving an investigational device or dictating care pathways at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred with intermediate likelihood of obstructive CAD with an Updated Diamond-Forrester (UDF) risk score 20-80% with symptomatic, suspected CAD
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Pontone, MD, Principal Investigator — Centro Cardiologico Monzino; Pamela Douglas, MD, Principal Investigator — Duke University; Bernard de Bruyne, MD, PHD, Principal Investigator — Cardiovascular Center Aalst; Mark Hlatky, MD, Principal Investigator — Stanford University
Locations (15):
- United States (3):
  - HeartFlow, Inc, Redwood City, California
  - Stanford University, Stanford, California
  - Duke University Clinical Research Institution, Durham, North Carolina
- Austria (2):
  - LKH-GRAZ-West - Department of Cardiology, Graz
  - Innsbruck Medical University, Department of Radiology II, Innsbruck
- Cardiovascular Center Aalst, Aalst, Belgium
- Aarhus University Hospital Skejby, Aarhus, Denmark
- France (2):
  - CHU Brest - Hopital de Cardiologie, Brest
  - Cardiovascular Hospital -Interventional Cardiology Dept, Hospices Civils de Lyon and Claude Bernard University France, Lyon
- Germany (3):
  - Heart Center Leipzig GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Deutsches Herzzentrum München - ISAResearch Centre, Munich
- Centro Cardiologico Monzino, Milan, Italy
- United Kingdom (2):
  - Freeman Hospital - Therapeutics & Cardiac Research Team, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Douglas PS, De Bruyne B, Pontone G, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C, Hlatky MA; PLATFORM Investigators. 1-Year Outcomes of FFRCT-Guided Care in Patients With Suspected Coronary Disease: The PLATFORM Study. J Am Coll Cardiol. 2016 Aug 2;68(5):435-445. doi: 10.1016/j.jacc.2016.05.057. PMID 27470449
- [Derived] Hlatky MA, De Bruyne B, Pontone G, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Wilk A, Wang F, Rogers C, Douglas PS; PLATFORM Investigators. Quality-of-Life and Economic Outcomes of Assessing Fractional Flow Reserve With Computed Tomography Angiography: PLATFORM. J Am Coll Cardiol. 2015 Dec 1;66(21):2315-2323. doi: 10.1016/j.jacc.2015.09.051. Epub 2015 Oct 14. PMID 26475205
- See also: 1-Year Outcomes of FFRCT-Guided Care in Patients With Suspected Coronary Disease: The PLATFORM Study — https://doi.org/10.1016/j.jacc.2016.05.057
- See also: Quality-of-Life and Economic Outcomes of Assessing Fractional Flow Reserve With Computed Tomography Angiography: PLATFORM — https://doi.org/10.1016/j.jacc.2015.09.051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be referred for non-invasive and/or invasive testing and evaluation. Prior to treatment of each subject considered for percutaneous coronary intervention (PCI) and/or coronary artery bypass grafting (CABG), the investigator and the institution's heart team will review clinical data and results of the diagnostic tests to recommend a treatment strategy, according to the institution's standard practice.
Pre-assignment Details: Patients were eligible for enrollment if they were symptomatic, had an intermediate likelihood of CAD, did not have an established diagnosis of CAD, and were referred for clinically indicated testing to evaluate CAD. Patients referred for noninvasive testing were enrolled in a separate stratum than patients referred for invasive testing. The choice to refer the patient for invasive testing rather than noninvasive testing was made by the local clinicians before enrollment in the study.
Groups:
- Non-invasive (Cohort 2) Usual Care: (Cohort 2) Subjects will be referred for non-invasive and/or invasive testing and evaluation. Prior to treatment of subjects considered for PCI and/or CABG, the investigator and the institution's heart team will review the results of all available diagnostic tests, including cCTA and FFRCT, and will recommend a treatment strategy accordingly.
- Non-invasive Cohort (Cohort 2) FFRCT; Invasive Cohort (Cohort 1) FFRCT: The second cohort of patients, enrolled after completion of the enrollment of the first cohort, was evaluated by CTA, with determination of FFRCT when a lesion of $30% stenosis was detected, or the patient was referred to invasive angiography.
- Invasive Cohort (Cohort 1) Usual Care: (Cohort 1) of the study is an observational evaluation of resource utilization and outcomes based on standard practice for diagnosis and treatment of subjects with symptomatic suspected CAD and intermediate likelihood of obstructive CAD.
Period: Overall Study
Arm/Group | Non-invasive (Cohort 2) Usual Care | Non-invasive Cohort (Cohort 2) FFRCT | Invasive Cohort (Cohort 1) Usual Care | Invasive Cohort (Cohort 1) FFRCT
Started | 100 | 104 | 187 | 193
Completed | 100 | 104 | 187 | 193
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Invasive Cohort (Cohort 1) Usual Care | Invasive Cohort (Cohort 1) FFRCT | Non-invasive (Cohort 2) Usual Care | Non-invasive Cohort (Cohort 2) FFRCT | Total
Number analyzed (Participants) | 187 | 193 | 100 | 104 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.36 (10.93) | 60.72 (10.20) | 57.91 (10.72) | 59.48 (9.33) | 60.86 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 34 | 44 | 231
  Male | 108 | 119 | 66 | 60 | 353
Diabetes [Count of Participants; unit: Participants] | 36 | 30 | 8 | 6 | 80
Current smoker [Count of Participants; unit: Participants] | 42 | 38 | 22 | 23 | 125
Hypertension [Count of Participants; unit: Participants] | 111 | 111 | 38 | 57 | 317
Hyperlipidemia [Count of Participants; unit: Participants] | 76 | 77 | 22 | 28 | 203
Atypical angina [Count of Participants; unit: Participants] | 122 | 142 | 91 | 80 | 435
Prior noninvasive testing [Count of Participants; unit: Participants] | 92 | 100 | 0 | 5 | 197
Pre-test probability of CAD [Count of Participants; unit: Participants] | 97 | 95 | 56 | 47 | 295

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Invasive Coronary Angiography
Description: The primary endpoint of the PLATFORM Study is 90 day (+30/-15 days) rate of coronary angiogram showing no stenosis > 50% in a vessel > 2.0 mm by Quantitative Coronary Angiography (QCA), or no invasively-measured FFR < 0.80 in a segment distal to a stenosis in a vessel > 2.0 mm by QCA between Cohort 1 and 2.
Time Frame: 90 Days from first test
Population: ICA - Invasive coronary angiography. Independent core laboratories performed quantitative coronary angiography.
Measure: Count of Participants; unit: Participants
Groups:
- Planned Invasive Test Usual Care Strategy (Cohort 1B): Cohort 1B consisted of subjects who were referred for ICA and were evaluated and treated according to standard practice.
- Planned Invasive Test FFRCT Guided Strategy (Cohort 2B): Cohort 2B also consisted of subjects who were referred for ICA, but instead had cCTA imaging, and then at the investigators discretion had FFRCT analysis performed.
Arm/Group | Planned Invasive Test Usual Care Strategy (Cohort 1B) | Planned Invasive Test FFRCT Guided Strategy (Cohort 2B)
Number analyzed (Participants) | 187 | 193
Participants | 137 | 24

2. Secondary Outcome: Number of MACE
Description: 90 days (+30/-30 days) Cohort 1 and Cohort 2 Major Adverse Coronary Event (MACE) rates, defined as:
  1. All cause death
  2. Non-fatal MI
  3. Unplanned hospitalization for acute coronary syndrome (ACS) leading to urgent revascularization
Time Frame: 90 days from first test
Population: The analysis population was defined as all subjects who were enrolled into the study. Safety was monitored throughout the study. The low number of MACE events made it impossible to analyze the powered secondary endpoint. None of the events were related to the FFRCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-invasive (Cohort 2) Usual Care | Non-invasive Cohort (Cohort 2) FFRCT | Invasive Cohort (Cohort 1) Usual Care | Invasive Cohort (Cohort 1) FFRCT
Number analyzed (Participants) | 100 | 104 | 187 | 193
Participants | 1 | 0 | 2 | 2

3. Secondary Outcome: Number of MACE or Vascular Complications
Description: 90 days (+30/-30 days) Major Adverse Coronary Event (MACE) rates, defined as: all cause death, non-fatal MI, unplanned hospitalization for acute coronary syndrome (ACS) leading to urgent revascularization and vascular complications (related to any coronary testing or procedure).This secondary endpoint compared the rates of MACE and vascular events across all subjects in Cohort 1 vs Cohort 2, Cohort 1A vs Cohort 2A and Cohort 1B vs Cohort 2B. The rates of MACE and vascular events were calculated by dividing the number of subjects with MACE and vascular events by the total number of subjects assigned to each analysis population.
Time Frame: 90 days from first test
Population: The analysis population was defined as all subjects who were enrolled into the study. It is important to note that none of the adverse events reported throughout the study were related to FFRCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-invasive (Cohort 2) Usual Care | Non-invasive Cohort (Cohort 2) FFRCT | Invasive Cohort (Cohort 1) Usual Care | Invasive Cohort (Cohort 1) FFRCT
Number analyzed (Participants) | 100 | 104 | 187 | 193
Participants | 0 | 1 | 2 | 7

4. Secondary Outcome: Number of Participants With Resource (CV Test Types Performed) Utilization at 90 Days
Description: Comparison of Resource utilization between cohort 1 and cohort 2 at 90 days (+/- 30 days):
  1. Non-invasive diagnostic tests
  2. Invasive diagnostic tests
  3. Coronary revascularization procedures
Time Frame: 90 days from first test
Measure: Count of Participants; unit: Participants
Groups:
- Non-invasive (Cohort 1A) Usual Care: Cohort 1A consisted of subjects presenting for their initial noninvasive test and were evaluated according to standard practice.
- Non-invasive Cohort (Cohort 2A) FFRCT: Cohort 2A also consisted of subjects presenting for their initial noninvasive test, but their first noninvasive test was cCTA with FFRCT analysis.
- Invasive Cohort (Cohort 1B) Usual Care: Cohort 1B consisted of subjects who were referred for ICA and were evaluated and treated according to standard practice.
- Invasive Cohort (Cohort 2B) FFRCT: Cohort 2B also consisted of subjects who were referred for ICA, but instead had cCTA imaging, and then at the investigators discretion had FFRCT analysis performed.
Arm/Group | Non-invasive (Cohort 1A) Usual Care | Non-invasive Cohort (Cohort 2A) FFRCT | Invasive Cohort (Cohort 1B) Usual Care | Invasive Cohort (Cohort 2B) FFRCT
Number analyzed (Participants) | 100 | 104 | 187 | 193
Participants
  ECG | 2 | 3 | 59 | 32
  Stress Echo | 2 | 0 | 7 | 6
  Nuclear/Stress MPI/CMR | 3 | 2 | 23 | 5
  cCTA without FFRCT | 8 | 2 | 21 | 12
  cCTA with FFRCT | 0 | 17 | 0 | 64
  IVUS, OCT, or FFR | 3 | 7 | 17 | 30
  ICA | 12 | 19 | 187 | 76
  PCI | 3 | 9 | 42 | 45
  CABG | 2 | 1 | 17 | 10

5. Secondary Outcome: Number of Participants With Medications Used by Type
Description: Comparison of medication use between cohort 1A, 1B and cohort 2A, 2B at 90 days (+/- 15 days)
Time Frame: at 90 days
Population: Values are the total number of patients who used particular medication (multiple medication types might be used per each patient)
Measure: Number; unit: participants (total count)
Arm/Group | Non-invasive (Cohort 1A) Usual Care | Non-invasive Cohort (Cohort 2A) FFRCT | Invasive Cohort (Cohort 1B) Usual Care | Invasive Cohort (Cohort 2B) FFRCT
Number analyzed (Participants) | 100 | 104 | 187 | 193
participants (total count)
  Aspirin | 29 | 45 | 115 | 90
  Statin | 24 | 29 | 83 | 77

ADVERSE EVENTS:
Time Frame: Clinical Outcomes at 1 Year
Description: All AEs were submitted to the independent clinical events committee (CEC) for review and adjudication. CEC adjudicated all MACE events in a blinded fashion using standard, prospectively determined definitions as described in Protocol.
Arm/Group | Non-invasive (Cohort 2) Usual Care | Non-invasive Cohort (Cohort 2) FFRCT | Invasive Cohort (Cohort 1) Usual Care | Invasive Cohort (Cohort 1) FFRCT
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/104 | 1/187 | 0/193
Serious Adverse Events (participants affected / at risk) | 2/100 | 1/104 | 6/187 | 9/193
Other Adverse Events (participants affected / at risk) | 6/100 | 13/104 | 137/187 | 24/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-invasive (Cohort 2) Usual Care (N=100) | Non-invasive Cohort (Cohort 2) FFRCT (N=104) | Invasive Cohort (Cohort 1) Usual Care (N=187) | Invasive Cohort (Cohort 1) FFRCT (N=193)
All-cause death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nonfatal MI (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hospitalization with urgent revascularization (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MACE or vascular complications (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-invasive (Cohort 2) Usual Care (N=100) | Non-invasive Cohort (Cohort 2) FFRCT (N=104) | Invasive Cohort (Cohort 1) Usual Care (N=187) | Invasive Cohort (Cohort 1) FFRCT (N=193)
Invasive catheterization without obstructive CAD (Cardiac disorders) | 6 (100) | 13 (104) | 137 (187) | 24 (193) — CAD - coronary artery disease. Obstructive CAD determined as 20%-80% stenosis by core lab quantitative coronary angiography (at 90 days).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less